CLINICAL TRIAL: NCT07347015
Title: Impact Evaluation of a Prescription Search Support (PSS) for Antimicrobials Using a Stepped-Wedge Cluster Randomized Design in Belgian Primary Care
Brief Title: Prescription Support System for Antimicrobial Use in Belgian Primary Care
Acronym: PaSSo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: National Institute for Health and Disability Insurance (RIZIV-INAMI) (Unknown); INTEGO - Flemish General Practice Morbidity Registry (KU Leuven) (Unknown); SMALS (Unknown)
Responsible Party: Principal Investigator, Jan Verbakel, Prof. Dr. Jan Y. Verbakel, KU Leuven
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: MP037810; MP037810 (Other: KU Leuven - Educational Review Board (OBC))
Record Dates: First submitted 2025-12-23; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Infectious Diseases
Keywords: Antimicrobial Stewardship; Primary Care; Clinical Decision Support; Stepped-Wedge Cluster Randomized Trial; Antibiotics
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: This study uses a stepped-wedge cluster randomized design to evaluate the implementation of a Prescription Support System (PSS) in Belgian primary care. All participating general practices start in a control condition and transition once to the intervention condition in four predefined steps over a nine-month period. Each step lasts three months. Practices contribute data during both control and intervention periods, allowing within- and between-cluster comparisons while accounting for time effects.
  Primary and secondary outcomes are based on routinely collected indicators from the Belgian Antibiotic Barometer. Analyses assess changes in antibiotic prescribing over time and compare practices by intensity of PSS use, derived from application log files. A process evaluation will be embedded, consisting of semi-structured interviews using a topic guide and log file analysis to assess implementation fidelity, reach and mechanisms of impact.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Usual Care (No Intervention): In the control arm, general practices will provide usual care, left at the discretion of the treating general practitioner.
  Apart from the general information or training session attended by all participating physicians prior to recruitment and randomization, practices in the control arm will not receive access to the Prescription Support System (PSS) or any additional decision support tools.
  General practitioners in the control arm are expected (but not forced) to follow the Belgian guidelines for antimicrobial prescribing, as described in the BAPCOC national guidelines.
- Intervention: access to PSS (Active Comparator): Prescription Support System (PSS) Providing guideline-based recommendations for antimicrobial prescribing in ambulatory care.
  Interventions: Other: Prescription Support System (PSS)

INTERVENTIONS:
Other: Prescription Support System (PSS) — General practices in this arm have access to the Prescription Support System (PSS), a digital clinical decision support tool integrated into the electronic health record that provides guideline-based recommendations for antimicrobial prescribing in ambulatory care. The PSS presents recommendations derived from the Belgian BAPCOC guidelines using a structured decision-tree format. During eligible consultations, the PSS can be consulted by the general practitioner to support clinical decision-making regarding antibiotic prescribing. The tool provides information on recommended antibiotic choice, dosage, and duration, as well as guidance on situations in which antibiotic treatment is not indicated. Practices transition to this arm according to the stepped-wedge design and retain access to the PSS for the duration of the study.
  Other Names: Clinical decision support system (CDSS)
  Arms: Intervention: access to PSS

SUMMARY:
Inappropriate antibiotic prescribing in primary care remains an important contributor to antimicrobial resistance. Despite the availability of evidence-based clinical guidelines, antibiotics are still frequently prescribed for self-limiting infections. Digital clinical decision support tools may help general practitioners (GPs) align prescribing decisions with guideline recommendations during patient consultations.

This study evaluates the impact of a digital Prescription Support System (PSS) designed to support antimicrobial prescribing in Belgian primary care. The PSS provides guideline-based recommendations derived from the Belgian BAPCOC guidelines for common infections in ambulatory care. Recommendations are presented through a user-friendly decision tree that is integrated into existing electronic health record systems and can be consulted during routine care.

The study is embedded within the national implementation strategy of the PSS coordinated by the National Institute for Health and Disability Insurance (RIZIV-INAMI). A stepped-wedge cluster randomized design is used, in which participating general practices transition sequentially from usual care to access to the PSS over four predefined implementation steps. This approach ensures that all participating practices eventually receive access to the system while allowing comparisons over time.

The primary objective is to assess whether implementation of the PSS is associated with changes in antibiotic prescribing in Belgian general practice. Prescribing outcomes are measured using routinely collected indicators from the Belgian Antibiotic Barometer, including overall antibiotic prescribing rates and the use of broad- versus narrow-spectrum antibiotics. Secondary objectives include assessing the usability and acceptability of the PSS among clinicians and identifying factors that influence its adoption in daily practice. The study will also monitor potential unintended consequences, such as changes in workflow or concerns about underprescribing.

Findings from this study will inform future decisions regarding further optimization and wider implementation of the PSS in Belgian primary care.

DETAILED DESCRIPTION:
Inappropriate antibiotic prescribing in primary care contributes to the development of antimicrobial resistance. Despite guidelines and public health efforts, overprescribing remains prevalent, especially for self-limiting infections which often resolve without antibiotic treatment. Digital tools such as a Prescription Search Support (PSS) may aid general practitioners (GPs) in making more informed prescribing decisions.

This implementation project builds upon a previously conducted mixed-methods implementation study evaluating the usability of a PSS, which was approved by the Ethical Review Board UZ KU Leuven (Onderwijs-Begeleidingscommissie) on 27 September 2024 (MP031770).

The PSS under study contains the current recommendations for the proper use of antimicrobial agents for common infections in ambulatory care in Belgium. In other words, it represents the BAPCOC guidelines in a digital and user-friendly environment, by using a decision tree. Advice for the following diagnoses (ICPC-2 codes) is included in the PSS: sore throat (R21, R74), pertussis (R71), common cold (R74), acute rhinosinusitis (R75), acute bronchitis / bronchiolitis (R78), influenza (R80), pneumonia (R81), ear pain (H01), otorrhea (H04), acute otitis media (H71), acute epiglottitis (R77), acute exacerbations of chronic obstructive pulmonary disease, aspiration pneumonia (R81), laryngitis stridulosa (R77), acute cystitis (U71), acute prostatitis (Y73), acute pyelonephritis (U70), acute vulvovaginitis (X84), asymptomatic bacteriuria, epididymo-orchitis (Y74), genital herpes (Y72, X90), partner treatment and treatment of asymptomatic sexually transmitted infections, pelvic inflammatory disease (X74), syphilis (X70, Y70), and urethritis (U72).

This PSS was developed as part of the Belgian National Action Plan on AMR by the Federal Public Service Health, Food Chain Safety and Environment and the National Institute for Health and Disability Insurance (NIHDI; RIZIV-INAMI), in collaboration with various experts and stakeholders, including physicians, infectiologists, hygienists, policymakers, guideline developers, and software developers. The company Smals, under instruction of RIZIV-INAMI, developed the software for this application in close collaboration with the RIZIV-INAMI working group. Guideline recommendations regarding appropriate prescribing of antimicrobials in ambulatory care were converted into decision rules, which serve as the knowledge source for the PSS.

Digital education offers several advantages, such as easy access without time or location constraints, varying possible forms and levels, and the ability to disseminate evidence on a large scale. Previous research has shown that standalone web- or smartphone-based applications in this context have the potential to increase physicians' knowledge of antimicrobials and guideline recommendations, potentially improving guideline adherence.

In Belgium, antibiotic use in ambulatory care is closely monitored through the Antibiotic Barometer, a national surveillance system coordinated by the Academic Centre of General Practice of KU Leuven and financed by the National Institute for Health and Disability Insurance (RIZIV-INAMI). The Antibiotic Barometer was approved by the Sociaal-maatschappelijke Ethische Commissie (SMEC; G-2023-6352) and provides quarterly feedback to general practices based on routine health insurance claims data.

This study evaluates the implementation and impact of the PSS in routine Belgian primary care using a stepped-wedge cluster randomized trial design. Participating general practices are recruited to ensure broad representation across Belgian primary care. General practices constitute the unit of randomization and are randomly allocated to one of four predefined implementation steps. All practices start in a control condition without access to the PSS and transition once to the intervention condition according to their assigned step. Each implementation step lasts three months, after which practices retain access to the PSS for the remainder of the study period. By the end of the study, all participating practices will have received access to the intervention.

Data for this study are derived from routine sources and handled within the secure data infrastructure of KU Leuven. Prescribing data obtained via the Antibiotic Barometer are aggregated and pseudonymized at practice level prior to analysis, ensuring that individual patients cannot be identified. Data linkage, storage, and analysis are conducted in accordance with applicable data protection regulations. Quantitative and qualitative analyses are used to evaluate both the effectiveness and implementation of the PSS in real-world primary care. Findings from this study will inform future policy decisions regarding national rollout, optimization, and long-term integration of the PSS within Belgian antimicrobial stewardship strategies.

ELIGIBILITY:
Inclusion Criteria:

* General practices in Belgium using compatible EHR systems.
* Willingness to use and activate the PSS by giving consent.
* Agreement to participate in the study, provided signed informed consent form is in place.

Exclusion Criteria:

* Practices using an EHR system that solely allows a single sign-on to the standalone PSS.
* Practices already using a similar PSS or participating in overlapping projects.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-21 (Estimated); Primary Completion 2026-12-21 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Antibiotic Prescribing Rate in General Practice | Measured quarterly from baseline until study completion (up to 12 months per practice).
  To evaluate whether the PSS reduces antibiotic prescribing rates in Belgian general practice. The project will assess whether implementation of the PSS tool leads to improvements in specific prescribing indicators as monitored by the Belgian Antibiotic Barometer (AB Barometer). These include total antibiotic prescribing rate and use of broad- versus narrow-spectrum antibiotics.

SECONDARY OUTCOMES:
Intensity of PSS use | Measured during the intervention period from each practice's transition to the PSS arm until study completion (up to 12 months).
  PSS usage intensity at practice level derived from application log files (e.g., frequency of access/consultations and categorization into high, medium, or no use during the intervention period), reflecting the overall level of exposure to the PSS.
Usability and acceptability of the PSS - clinician reported | Assessed after transition to the intervention group, during the final 6 months of the study period.
  To assess the usability of the Prescription Support System (PSS) among general practitioners in routine clinical practice. Usability will be explored through semi-structured interviews with clinicians. The evaluation will examine clinicians' experiences with the PSS, perceived usefulness, ease of use, and integration into workflow, and factors influencing adoption, sustained use, and perceived impact on prescribing decisions.
Usability and acceptability of the PSS - system usage | Assessed during the intervention period from each practice's transition to the PSS arm until study completion (up to 12 months).
  Usability of the Prescription Support System (PSS) will also be assessed using system usage data derived from application log files, including patterns of use and interaction with the PSS during routine clinical practice, focusing on how the system is used rather than how often it is accessed.
Potential Unintended Consequences of PSS Implementation - clinician reported | Assessed after transition to the intervention group, during the final 6 months of the study period.
  To monitor potential unintended consequences associated with implementation of the Prescription Support System (PSS), including perceived workflow disruption. These outcomes will be explored using qualitative information obtained through semi-structured interviews with clinicians.
Potential Unintended Consequences of PSS Implementation - system usage | Measured quarterly from baseline until study completion (up to 12 months)
  To monitor potential unintended consequences associated with implementation of the Prescription Support System (PSS), including signals of underprescribing and changes in prescribing patterns. These outcomes will be explored using routinely collected prescribing indicators from the Belgian Antibiotic Barometer.

CONTACTS AND LOCATIONS:
Locations (1):
- GPs associated with KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data from this trial will not be published in the public domain. Deidentified participant data is available for further analyses. Requests for data, with justification, should be sent to Jan Verbakel (jan.verbakel@kuleuven.be). The trial protocol is available online for an indefinite period.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study protocol is published and accessible. SAP, CSR, ICF and analytical code will be available after publishing the results in a medical journal. Individual patient data from this trial will not be published in the public domain.
Access Criteria: Individual patient data from this trial will not be published in the public domain. Deidentified participant data is available for further analyses. Requests for data, with justification, should be sent to Jan Verbakel (jan.verbakel@kuleuven.be). The trial protocol is available online for an indefinite period.

REFERENCES:
- [Background] Madar R, Ugon A, Ivankovic D, Tsopra R. A Web Interface for Antibiotic Prescription Recommendations in Primary Care: User-Centered Design Approach. J Med Internet Res. 2021 Jun 11;23(6):e25741. doi: 10.2196/25741. PMID 34114958
- [Background] Delory T, Jeanmougin P, Lariven S, Aubert JP, Peiffer-Smadja N, Boelle PY, Bouvet E, Lescure FX, Le Bel J. A computerized decision support system (CDSS) for antibiotic prescription in primary care-Antibioclic: implementation, adoption and sustainable use in the era of extended antimicrobial resistance. J Antimicrob Chemother. 2020 Aug 1;75(8):2353-2362. doi: 10.1093/jac/dkaa167. PMID 32357226
- [Background] Helou RI, Foudraine DE, Catho G, Peyravi Latif A, Verkaik NJ, Verbon A. Use of stewardship smartphone applications by physicians and prescribing of antimicrobials in hospitals: A systematic review. PLoS One. 2020 Sep 29;15(9):e0239751. doi: 10.1371/journal.pone.0239751. eCollection 2020. PMID 32991591
- [Background] Fralick M, Haj R, Hirpara D, Wong K, Muller M, Matukas L, Bartlett J, Leung E, Taggart L. Can a smartphone app improve medical trainees' knowledge of antibiotics? Int J Med Educ. 2017 Nov 30;8:416-420. doi: 10.5116/ijme.5a11.8422. PMID 29200402
- [Background] Kyaw BM, Tudor Car L, van Galen LS, van Agtmael MA, Costelloe CE, Ajuebor O, Campbell J, Car J. Health Professions Digital Education on Antibiotic Management: Systematic Review and Meta-Analysis by the Digital Health Education Collaboration. J Med Internet Res. 2019 Sep 12;21(9):e14984. doi: 10.2196/14984. PMID 31516125
- [Background] 1. BAPCOC - Belgische Gids voor Anti-Infectieuze Behandeling in de Ambulante Praktijk 2022. Available from: https://www.bcfi.be/nl/chapters/12?frag=8000010. Accessed 11 July 2024.